CLINICAL TRIAL: NCT05885724
Title: Novel Targetable BIOmarkers in ANorexia NervosA - BIOANNA
Brief Title: Novel Targetable BIOmarkers in ANorexia NervosA
Acronym: BIOANNA
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-00513, kt23Timper2
Record Dates: First submitted 2023-05-22; First posted 2023-06-02 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Anorexia Nervosa; Anorexia Nervosa Restricting Type
Keywords: exercising subtype; non-exercising subtype; Neurofilament light chain; Glial fibrillary acidic protein; Growth Differentiation Factor-15
MeSH Terms: conditions — Anorexia Nervosa; Charcot-Marie-Tooth disease, Type 1F

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The overall aim of this present study is to evaluate Growth Differentiation Factor-15 (GDF-15) and inflammatory cytokines as a possible novel and readily treatable target for the successful therapy of Anorexia Nervosa (AN). Therefore, GDF-15, neuronal and glial damage markers such as Neurofilament light chain (Nfl) and Glial fibrillary acidic protein (GFAP) and cytokines (such as Tumor necrosis factor alpha (TNF-α), Interleukin-6 (IL-6), and Interleukin 1β (IL-1β) levels will be assessed in the serum as well as in the cerebrospinal fluid of patients with diagnosed restrictive AN with and without exercising behavior compared to sex- and age-matched healthy controls to consolidate previous findings and to identify the main site of production of GDF-15 and cytokines in AN.

DETAILED DESCRIPTION:
In addition, assessment of body composition via Dual Energy X-ray Absorptiometry (DEXA )scans and of energy expenditure via indirect calorimetry, respectively, will allow us to correlate GDF-15, Nfl and GFAP and cytokine levels with lean and fat mass measures as well as with energy expenditure, respectively, of AN patients and the matched controls. Overall, this will allow us to comprehensively evaluate GDF-15 and cytokines as possible novel targets for the treatment of AN and to set the basis for a follow up study using available neutralizing antibodies or inhibitors against GDF-15 and the respective cytokines for the treatment of patients with AN, respectively. This will also allow for a more tailored, individualized treatment approach of AN in the future. Our findings will hopefully challenge the viewpoint that AN is a condition which can be controlled by the individual but demonstrate that AN is a biological disease that should be treated by targeting the right biological players in addition to psychiatric treatment.

ELIGIBILITY:
N=8 adult male and female patients with confirmed diagnosis of anorexia nervosa restrictive type, non-exercising subtype

Inclusion criteria:

* Age 18-60 years
* Written informed consent
* BMI 10-16 kg/m2

N=8 adult male and female patients with confirmed diagnosis of anorexia nervosa restrictive type, exercising subtype will be included in this study.

Inclusion criteria:

* Age 18-60 years
* Written informed consent
* BMI 10-16 kg/m2

N=16 control participants, sex- and age-matched to the individual anorexia nervosa patients.

Inclusion criteria:

* Age 18-60 years
* Written informed consent
* BMI 19-24.9 kg/m2

Exclusion Criteria:

* Use of antibiotics within the last 31 days
* Current illicit drug abuse including daily marijuana or CBD (cannabidiol) consumption (≤ 24 g of alcohol per day allowed)
* Any kind of severe chronic disease other than AN (e.g. active cancer disease)
* Severe renal impairment (e.g. estimated glomerular filtration rate <30 ml/min/m2) if resulting from another disease than AN
* Known liver cirrhosis or other severe liver impairment if resulting from another disease than AN
* Acute upper respiratory tract infection within the last 31 days
* Uncontrolled dysthyroidism
* Uncontrolled hypertension
* Current pregnancy/lactation or current treatment for in vitro fertilization
* Inability to understand the study information, to sign the consent form and to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients with confirmed diagnosis of AN will be recruited via the anorexia outpatient clinic of the Endocrinology Department, University Hospital Basel, headed by Prof. Dr. Katharina Timper and via advertisement. Healthy sex- and age (+/- 3 years of age difference) control participants will be recruited at the medical and endocrinology outpatient clinic of the University Hospital of Basel and via advertisement.
Sampling Method: Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Growth Differentiation Factor-15 (GDF-15) (pg/ml) level in the plasma | one time assessment 3 weeks after screening
  Comparison of GDF-15 (pg/ml) level in the plasma of AN patients and normal-weight controls Blood in overnight-fasted study participants will be taken from a cubital vein and analyzed for GDF-15 (pg/ml)
Growth Differentiation Factor-15 (GDF-15) (pg/ml) level in the cerebrospinal fluids | one time assessment 3 weeks after screening
  Comparison of GDF-15 level in the cerebrospinal fluids of AN patients and normal-weight controls. CSF will be analysed only from patients who undergo a liquor puncture as part of their clinical assessment and consent to having taken an extra 5ml. Cerebrospinal fluid (CSF) will then be analysed for GDF-15 (pg/ml)

CONTACTS AND LOCATIONS:
Overall Officials: Katharina Timper, Prof., Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Switzerland